CLINICAL TRIAL: NCT00823524
Title: Donor NK Cell Infusion for Progression/Recurrence of Underlying Malignant Disorders After HLA-haploidentical HCT - a Phase 1-2 Study
Brief Title: Donor Natural Killer Cells After Donor Stem Cell Transplant in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Korea Research Institute of Bioscience & Biotechnology (Other Government)
Responsible Party: Principal Investigator, Kyoo-Hyung Lee, Professor of Internal Medicine, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000632275; AMC-UUCM-2008-0383
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Brain and Central Nervous System Tumors; Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Lymphoproliferative Disorder; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: accelerated phase chronic myelogenous leukemia; acute undifferentiated leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL1 negative; blastic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; mast cell leukemia; meningeal chronic myelogenous leukemia; progressive hairy cell leukemia, initial treatment; prolymphocytic leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult T-cell leukemia/lymphoma; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage III adult T-cell leukemia/lymphoma; stage III chronic lymphocytic leukemia; stage IV adult T-cell leukemia/lymphoma; stage IV chronic lymphocytic leukemia; T-cell large granular lymphocyte leukemia; adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; splenic marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage III mycosis fungoides/Sezary syndrome; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage IV mycosis fungoides/Sezary syndrome; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; intraocular lymphoma; primary central nervous system non-Hodgkin lymphoma; primary central nervous system Hodgkin lymphoma; post-transplant lymphoproliferative disorder; chronic eosinophilic leukemia; chronic neutrophilic leukemia; primary myelofibrosis; essential thrombocythemia; polycythemia vera; extramedullary plasmacytoma; isolated plasmacytoma of bone; stage II multiple myeloma; stage III multiple myeloma; primary systemic amyloidosis; refractory multiple myeloma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; cutaneous B-cell non-Hodgkin lymphoma; Waldenström macroglobulinemia; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Central Nervous System Neoplasms; Myeloproliferative Disorders; Leukemia; Lymphoma; Lymphoproliferative Disorders; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Mast-Cell; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Intraocular Lymphoma; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Primary Myelofibrosis; Thrombocythemia, Essential; Polycythemia Vera; Immunoglobulin Light-chain Amyloidosis; Waldenstrom Macroglobulinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- donor NK cell infusion (Experimental): give patients donor-derived NK cells 2 to 3 weeks after HLA-haploidentical hematopoietic cell transplantation
  Interventions: Biological: donor natural killer cell infusion

INTERVENTIONS:
Biological: donor natural killer cell infusion — give patients donor-derived NK cells 2 to 3 weeks after HLA-haploidentical hematopoietic cell transplantation

SUMMARY:
RATIONALE: Giving an infusion of natural killer cells from a donor after a donor stem cell transplant may help kill any remaining cancer cells after the transplant.

PURPOSE: This phase I/II trial is studying the side effects and best dose of donor natural killer cells when given after a donor stem cell transplant in treating patients with advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the safety of donor natural killer (NK) cell infusion after HLA-mismatched/haploidentical allogeneic hematopoietic stem cell transplantation from a familial donor in patients with advanced malignant disorders.
* To determine the maximum number of donor NK cells that can be safely given to these patients.

Secondary

* To assess the clinical efficacy donor NK cell infusion, in terms of tumor response, response duration, and survival, in patients with progressive or recurrent malignant disorders.

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

* Phase I: Patients receive an infusion of donor natural killer (NK) cells on days 18 and 21.
* Phase II: Patients receive an infusion of donor NK cells on days 14 and 21. After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a malignant disorder (hematologic malignancies or solid tumors)

  * Advanced disease
* Has undergone prior allogeneic hematopoietic stem cell transplantation (HSCT) from an HLA-mismatched/haploidentical familial donor
* Progressive or recurrent disease, as defined by any of the following (phase II):

  * Peripheral blood blast > 20% with bone marrow aspirate showing > 5% leukemic cells (in patients with acute leukemia)
  * Detection of metaphases in the marrow with the same clonal cytogenetic abnormalities as identified before HSCT (or by FISH markers, if appropriate) (in patients with acute leukemia or high-risk myelodysplastic syndromes [MDS])
  * Persistent cytopenia with bone marrow aspirate showing various degrees of dysplasia involving ≥ 1 cell lineage (in patients with high-risk MDS)
  * Enlargement of pre-existing measurable lesions by 20% according to RECIST criteria (in patients with solid tumors or lymphoma)
  * Appearance of new metastatic lesions, including pleural effusion or ascites, radiologically typical for metastases or confirmed as such by cytology (in patients with solid tumors or lymphoma)
* Measurable disease (phase II)

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Total bilirubin < 3.0 mg/dL
* AST < 5 times upper limit of normal
* Creatinine < 3 mg/dL
* Not pregnant or nursing
* No clinically evident cardiac or pulmonary failure

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Safety | 15 days to 1 year after transplantation
  Safety will be evaluation in terms of transplantation outcomes as well as side effects of donor NK cell infusion

SECONDARY OUTCOMES:
Clinical efficacy of donor NK cell infusion, in terms of tumor response, response duration, and survival | 15 days to 1 year
  achievement of CR of underlying disease, CR duration

CONTACTS AND LOCATIONS:
Overall Officials: Kyoo H. Lee, MD, Principal Investigator — Asan Medical Center
Locations (1):
- University of Ulsan, Asan Medical Center, Seoul, South Korea